NCT04287517 10.12.2019

# Efficacy of Capacitive-Resistive Therapy on the Treatment of Myofascial Pain

Informed Consent Form

NCT04287517 10.12.2019

## **Informed Consent Form**

This Informed Consent Form was prepared to invite adult individuals to study of "Efficacy of Capacitive-Resistive Therapy on the Treatment of Myofascial Pain".

Name and Surname of the Researcher:

Name and Surname of the Assistant Researcher:

*Name of the institution that will conduct the research:* 

#### Introduction

You have been invited to participate in the study called " *Efficacy of Capacitive-Resistive Therapy on the Treatment of Myofascial Pain*". Before accepting to take part in this study, you need to understand what purpose and how the study will be done and make your decision about whether or not to participate freely after this information. The information that I will give to you orally about the research will be presented to you in writing in the next section. Please read this document carefully, ask for clear answers to your questions. The last section in this document is about approval procedures. If you agree to participate in the research, please sign this section. If you have obstacles to reading and writing, you will be asked to approve this document under the supervision of a witness and your fingerprint will be taken if necessary.

# Information About Study

Myofascial pain syndrome (MPS) is a painful musculoskeletal condition affecting the individuals' daily life presenting with muscle spasm, referred pain patterns, stiffness, restricted range of motion caused by trigger points. Capacitive-resistive diathermy therapy heats deep tissues by transferring energy through radiofrequency waves. Currently, although this modality is used to treat various acute or chronic musculoskeletal disorders, there is no specific data about myofascial trigger points in the literature. We aimed to evaluate the efficacy of capacitive-resistive diathermy on the myofascial trigger point of neck/upper trapezius muscle area compared with the sham intervention of capacitive-resistive diathermy.

Capacitive-resistive therapy will be applied to the trigger points on the trapezius muscle in the neck muscle group in this study. We will examine individual's pain, range of motion, and quality of daily life. The patient's evaluations will be made using VAS (Visual Analog Scale), analog algometer, digital inclinometer, NDI (Neck Disability Index) questionnaire, SF-36 (Short form 36 health scale) questionnaire. Detailed information will be given about how the application will be done before all applications. Before the study, patients will be randomly divided into two groups, one group will be given capacitive-resistive therapy and exercise, the other group will be given sham (placebo) capacitive-resistive therapy and exercise. Patients will be treated in the sports medicine clinic with a physiotherapist for 10 days in 3 weeks. The above evaluations and surveys will be done before and after treatment under supervision of specialist and physiotherapist.

NCT04287517 10.12.2019

### Information on Volunteer's Rights

The above information about this research was conveyed to me by stating that a research will be conducted by the specialist on the " Efficacy of Capacitive-Resistive Therapy on the Treatment of Myofascial Pain". After this briefing, I was invited to participate in such a research as a "volunteer". If I participate in this research, I have been assured that the information that I have to keep with the doctor will be protected confidentially and with great care and respect. I have been given sufficient confidence that my personal information will be carefully protected during the use of research results for educational and scientific purposes. I can withdraw from the research without showing any reason during the conduct of the research. I can also be excluded from the research by the researcher, provided that my medical condition is not harmed. I do not assume any monetary responsibility for the expenditures for the research. I will not be paid a fee (it should be stated separately if some payments will be made, such as compensating for travel money, food, or lagging work). Necessary assurance was provided that any medical intervention would be provided if any health problems that may arise from the research application, whether direct or indirect, arise. I will not be under a monetary burden regarding these medical interventions. When I encounter a health problem during the research; at any time, I know that I can call the specialist on 0090 212 414 24 42. I do not have to participate in this research and may not participate. I have not encountered compelling behavior in participating in the research. I also know that if I refuse to participate, this will not harm my medical care and my relationship with the doctor.

Name and Surname of the Volunteer:

Volunteer's Address and Phone Number:

Signature of the Volunteer:

Name and Surname of the Researcher:

Researcher's Address and Phone Number:

Signature of the Researcher:

Name and Surname of the Assistant Researcher:

Assistant Researcher's Address and Phone Number:

Signature of the Assistant Researcher: